CLINICAL TRIAL: NCT00975780
Title: A Randomized Controlled Trial to Reduce Pneumonia in Nursing Home Residents
Brief Title: A Trial to Reduce Pneumonia in Nursing Home Residents
Acronym: PRIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0609001783; R01AG030575 (NIH)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2014-01-21 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Pneumonia; Lower Respiratory Tract Infection
Keywords: Pneumonia; Lower respiratory tract infection; Lower respiratory tract infection other than pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enhanced oral care (Experimental)
  Interventions: Other: Enhanced Oral Care
- Usual care (Active Comparator): The usual oral care provided at the nursing home
  Interventions: Other: Usual oral care

INTERVENTIONS:
Other: Enhanced Oral Care — oral brushing plus oral chlorhexidine plus upright feeding positioning
  Arms: enhanced oral care
Other: Usual oral care — Usual oral care and feeding positioning
  Arms: Usual care

SUMMARY:
The purpose of this study is to test the effectiveness of an enhanced oral hygiene protocol in preventing pneumonia among nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

* long term care resident of nursing home
* residents age >65
* residents of nursing home for at least one month
* residents having at least one of two modifiable risk factors for pneumonia (i.e., impaired oral hygiene, swallowing difficulty)

Exclusion Criteria:

* residents housed in nursing home for short term rehabilitation
* residents who receive nourishment by tube feeding
* residents who have a life expectancy < 3 months
* residents who have been diagnosed with pneumonia within the previous 6 weeks
* residents who are currently using oral chlorhexidine
* residents who have previously been enrolled in the study
* residents, or their designated proxies, who are unwilling to give informed consent
* residents who have tracheostomy
* residents who are non-english speaking
* residents who the administrator leadership of the home felt were not appropriate for the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 834 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent J Quagliarello, MD, Principal Investigator — Yale University; Mary Tinetti, MD, Study Director — Yale University; Manisha Juthani-Mehta, MD, Study Director — Yale University; Peter Peduzzi, PhD, Study Director — Yale University; Dorothy Baker, PhD, Study Director — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Juthani-Mehta M, Van Ness PH, McGloin J, Argraves S, Chen S, Charpentier P, Miller L, Williams K, Wall D, Baker D, Tinetti M, Peduzzi P, Quagliarello VJ. A cluster-randomized controlled trial of a multicomponent intervention protocol for pneumonia prevention among nursing home elders. Clin Infect Dis. 2015 Mar 15;60(6):849-57. doi: 10.1093/cid/ciu935. Epub 2014 Dec 16. PMID 25520333

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: The usual oral care provided at the nursing home
  Usual oral care : Usual oral care and feeding positioning
- Enhanced Oral Care: Enhanced Oral Care : oral brushing plus oral chlorhexidine plus upright feeding positioning
Period: Allocation
Arm/Group | Usual Care | Enhanced Oral Care
Started | 400 | 434
Completed | 400 | 434
Not Completed | 0 | 0
Period: Follow Up
Arm/Group | Usual Care | Enhanced Oral Care
Started | 400 | 434
Completed | 298 | 277
Not Completed | 102 | 157
Not completed — Death | 88 | 122
Not completed — Facility Withdrawal | 7 | 23
Not completed — Discharged from Facility | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Oral Care: Study participants receiving 'Enhanced Oral Care' in the study
- Usual Oral Care: Study participants receiving 'Usual Oral Care' in the study.
- Total: Total of all reporting groups
Arm/Group | Enhanced Oral Care | Usual Oral Care | Total
Number analyzed (Participants) | 434 | 400 | 834
Age, Continuous [Mean (Standard Deviation); unit: years] | 86.5 (8.0) | 86.1 (8.3) | 86.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329 | 307 | 636
  Male | 105 | 93 | 198

OUTCOME MEASURES:

1. Primary Outcome: Pneumonia
Description: The number of participants that recorded a 'first pneumonia' during the 2.5 years timeframe.
Time Frame: 2.5 years
Measure: Number; unit: participants
Arm/Group | Enhanced Oral Care | Usual Oral Care
Number analyzed (Participants) | 434 | 400
participants | 119 | 94

2. Secondary Outcome: Lower Respiratory Tract Infection Other Than Pneumonia
Description: The number of participants that recorded a 'lower respiratory tract infection other than pneumonia' during the 2.5 years timeframe.
Time Frame: 2.5 years
Measure: Number; unit: participants
Arm/Group | Enhanced Oral Care | Usual Oral Care
Number analyzed (Participants) | 434 | 400
participants | 125 | 100

ADVERSE EVENTS:
Time Frame: Adverse events (both Serious and Other) were collected over the 2.5 year study period.
Arm/Group | Enhanced Oral Care | Usual Oral Care
Serious Adverse Events (participants affected / at risk) | 204/434 | 153/400
Other Adverse Events (participants affected / at risk) | 391/434 | 371/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Oral Care (N=434) | Usual Oral Care (N=400)
Urinary Tract Infection (Renal and urinary disorders) | 19 (23) | 13 (19)
Skin / Soft Tissue Event (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Eye Infection (Eye disorders) | 0 (0) | 2 (2)
Respiratory Difficulty (Respiratory, thoracic and mediastinal disorders) | 52 (74) | 37 (51)
Fall (General disorders) | 16 (19) | 20 (21) — Defined as a study participant falling down; the resulting injury leading to hospitalization.
Acute Renal Failure (Renal and urinary disorders) | 6 (8) | 3 (4)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastrointestinal Disturbance (Gastrointestinal disorders) | 20 (27) | 21 (26)
Abnormal Blood Glucose (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute Chest Pain/Coronary Syndrome (Cardiac disorders) | 2 (2) | 8 (8)
Altered Mental Status (Psychiatric disorders) | 33 (38) | 22 (27)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Blood Pressure Alteration (Vascular disorders) | 1 (1) | 2 (2)
Weight Loss (General disorders) | 0 (0) | 1 (1)
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fever (Infections and infestations) | 8 (10) | 6 (6)
Generalize Malaise (Psychiatric disorders) | 0 (0) | 1 (1)
Other (General disorders) | 38 (41) | 22 (28) — These Serious Adverse Events were those that led to hospitalization that were otherwise not specified. Given the characteristics of the study population (age, environment), hospitalization is not uncommon.
Unrelated and Unanticipated OTHER (General disorders) | 0 (0) | 2 (2) — Unrelated and unanticipated OTHER events deemed to be Serious Adverse Events.
Death (General disorders) | 125 (125) | 95 (95) — Death (unrelated to intervention)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Oral Care (N=434) | Usual Oral Care (N=400)
Urinary Tract Infection (Renal and urinary disorders) | 156 (270) | 130 (211)
Skin / Soft Tissue Event (Skin and subcutaneous tissue disorders) | 271 (880) | 217 (669)
Eye Infection (Eye disorders) | 81 (131) | 66 (84)
Respiratory Difficulty (Respiratory, thoracic and mediastinal disorders) | 238 (482) | 228 (449)
Fall (General disorders) | 143 (300) | 138 (277)
Gastrointestinal Disturbance (Gastrointestinal disorders) | 161 (347) | 115 (230)
Altered Mental Status (Psychiatric disorders) | 98 (184) | 66 (129)
Joint Pain (Musculoskeletal and connective tissue disorders) | 76 (118) | 64 (107)
Back Pain (Musculoskeletal and connective tissue disorders) | 36 (46) | 25 (36)
Oral Cavity Disturbance (General disorders) | 51 (57) | 55 (72)
Weight Loss (General disorders) | 36 (46) | 21 (22)
Headache (General disorders) | 33 (51) | 25 (36)
Leg Pain (Musculoskeletal and connective tissue disorders) | 23 (27) | 15 (24)
Fever (Infections and infestations) | 34 (43) | 22 (26)
Generalized Malaise (General disorders) | 31 (35) | 18 (31)

LIMITATIONS AND CAVEATS:
Participant flow and outcome information pertains to data collected through 10/25/2012- the official trial termination date.

Serious and Other Adverse Event information pertains to requested surveillance of subjects through 12/10/2012 per the NIA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes